CLINICAL TRIAL: NCT04521608
Title: Increasing Adherence to Pulmonary Rehabilitation After COPD Related Hospitalizations
Brief Title: Increasing Adherence to Pulmonary Rehabilitation After COPD Related Hospitalizations (Study 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-002453; R61HL142933 (NIH)
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention- Home Pulmonary Rehabilitation (Experimental): Participants enrolled in the intervention arm will be offered a Home-based pulmonary rehabilitation program with health coaching.
  Interventions: Behavioral: Intervention- Home-based Pulmonary Rehabilitation
- Control- Choice (No Intervention): This arm was the choice of Pulmonary Rehabilitation at a facility or Home-based pulmonary rehabilitation program with health coaching.

INTERVENTIONS:
Behavioral: Intervention- Home-based Pulmonary Rehabilitation — Home-based Pulmonary Rehabilitation (PR) with health coaching using a remote system that will allow patients to complete PR at home. The program involves upper and lower extremity exercises, self-report of symptoms (fatigue, breathlessness, physical activity and overall well-being).
  Arms: Intervention- Home Pulmonary Rehabilitation

SUMMARY:
This study is being done to test the comparative effectiveness of participating in a Pulmonary Rehabilitation Program at home using new technology and health coaching following dismissal from the hospital compared to the referral to a center based pulmonary rehabilitation that may include the choice of center based or telehealth.

DETAILED DESCRIPTION:
Despite proven benefits, the proportion of people with COPD who receive Pulmonary Rehabilitation (PR) is very small. The current model of a center-based PR program fails to address the needs of many patients with COPD. After the COVID epidemic, telehealth is an option for individuals referred to patients referred to center based rehabilitation.

The direct referral to home-based, unsupervised PR has been proposed as an alternative model to hospital-based programs and has been found to be safe and effective. The refined home-based PR program from the pilot portion of the study supported by a separate grant mechanism (R61HL142933/NCT03865329) will be tested in this second part randomized control study.

Subjects with a COPD-related hospitalization (exacerbation or pneumonia) will be randomized after hospital discharge to either home-based PR or Choice (referral to conventional center-based PR or home-based PR.

ELIGIBILITY:
Inclusion Criteria:

* COPD related hospitalization and eligible for PR
* Age 40+
* Confidence (score > 5 in a self-efficacy question (1-10 scale): how confident you feel to use this system on a daily basis)

Exclusion Criteria:

- Inability to walk (orthopedic-neurologic problems or confined to bed)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Health Partners Institute, Bloomington, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 296 participants were consented to the study. 2 participants were withdrawn from the study before assignment to groups.
Groups:
- Intervention- Home Pulmonary Rehabilitation: Participants enrolled in the intervention arm were offered a Home-based pulmonary rehabilitation program with health coaching.
  Intervention- Home-based Pulmonary Rehabilitation: Home-based Pulmonary Rehabilitation (PR) with health coaching using a remote system that allowed patients to complete PR at home. The program involved upper and lower extremity exercises, self-report of symptoms (fatigue, breathlessness, physical activity and overall well-being).
- Control- Choice: This arm received the standard of care which included the choice of PR at a facility or through telehealth. Center based PR involved attending a medical center gym where they could do exercises and receive disease specific education. Telehealth PR was delivered virtually through the computer or telephone.
Period: Overall Study
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice
Started | 147 | 147
Completed | 66 | 73
Not Completed | 81 | 74
Not completed — Death | 8 | 9
Not completed — Withdrawal by Subject | 25 | 18
Not completed — Disease Progression | 3 | 10
Not completed — Complicating Disease | 6 | 3
Not completed — Lost Contact | 25 | 27
Not completed — Ineligible | 1 | 0
Not completed — Refused Further Study Participation | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice | Total
Number analyzed (Participants) | 147 | 147 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.52 (8.99) | 70.39 (8.56) | 70.45 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 77 | 155
  Male | 69 | 70 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 142 | 138 | 280
  Unknown or Not Reported | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 4 | 11
  White | 138 | 141 | 279
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 147 | 147 | 294

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Pulmonary Rehabilitation (PR)
Description: The number of subjects who completed PR through 3 months
Time Frame: baseline; 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice
Number analyzed (Participants) | 147 | 147
Participants | 82 | 95

2. Primary Outcome: Change in Health Related Quality of Life as Measured by the Chronic Respiratory Questionnaire (CRQ).
Description: The Chronic Respiratory Questionnaire (CRQ) is a validated tool that is completed by participants at baseline and 3 months, measuring health-related quality of life. This questionnaire measures both physical and emotional aspects of chronic respiratory disease. We reported the difference between baseline and 3 months on the CRQ emotional summary scores (comprised of the summation of the mastery and emotional domains of CRQ divided by 2) and the physical summary score (comprised of the summation of the dyspnea and fatigue domains of the CRQ divided by 2). Summary scores as well as the original domains , all have a range of 1 to 7 points, with a higher number being a better health-related quality of life. 0.5 points is the minimal clinically important difference for this tool. Then, for the interpretation of CRQ results: a difference>0.5 is considered clinically meaningful
Time Frame: baseline; 3 months
Population: The results are presented as the difference between baseline and month 3 (end of the intervention). For the interpretation of CRQ results: a difference>0.5 is considered clinically meaningful
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice
Number analyzed (Participants) | 80 | 91
score on a scale
  CRQ Physical Summary Score | 0.37 [0.18 to 0.56] | 0.8 [0.59 to 1.01]
  CRQ Emotional Summary Score | 0.46 [0.24 to 0.69] | 0.6 [0.4 to 0.8]

3. Primary Outcome: Change in EuroQol (EQ-5D) Score
Description: The EuroQol (EQ-5D) is a 5-item questionnaire that assesses health-related quality of life over five different dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. It also includes a Visual Analogue Scale (VAS) for self-related heath. Each dimension uses a 5-level Likert scale (1 = no problems, 5 = extreme problems), ensuring nuanced data collection. The VAS ranges from 0 (worst imaginable health) to 100 (best imaginable health). Scores are calculated for each dimension with total scores ranging from 1 (no problems) to 5 (extreme problems), with higher scores indicating a worse outcome. The score from the VAS portion of the questionnaire ranges from 0 (worst imaginable health) to 100 (best imaginable health), with higher scores indicating a better outcome.
Time Frame: baseline; 3 months
Population: 1 subject in the intervention arm was not included in the analysis for the health today (VAS score) score of the questionnaire and 1 subject in the choice arm was not included in the analysis for the pain/discomfort score of the questionnaire as both subjects inadvertently skipped those sections of the questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice
Number analyzed (Participants) | 80 | 91
score on a scale
  Mobility | -0.28 [-0.49 to -0.06] | -0.23 [-0.42 to -0.04]
  Self Care | -0.22 [-0.43 to -0.02] | -0.08 [-0.19 to 0.04]
  Usual Activities | -0.25 [-0.44 to -0.06] | -0.16 [-0.36 to 0.03]
  Pain/Discomfort: number analyzed (Participants) | 80 | 90
  Pain/Discomfort | 0.06 [-0.11 to 0.24] | -0.24 [-0.4 to -0.09]
  Anxiety/Depression | -0.09 [-0.26 to 0.09] | -0.21 [-0.39 to -0.03]
  Health Today (VAS Score): number analyzed (Participants) | 79 | 91
  Health Today (VAS Score) | 3.27 [-1.56 to 8.1] | 8.16 [4.15 to 12.18]

4. Secondary Outcome: Number of Subjects Who Visited the Emergency Department
Description: The number of subjects who had at least one Emergency Department visit from baseline to 3 months.
Time Frame: baseline to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice
Number analyzed (Participants) | 82 | 95
Participants | 18 | 24

5. Secondary Outcome: Number of Subjects Who Had a Hospitalization
Description: The number of subjects who had at least one hospitalization from baseline to 3 months.
Time Frame: baseline; 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice
Number analyzed (Participants) | 82 | 95
Participants | 23 | 21

6. Secondary Outcome: Change in Self-Management Ability Scale
Description: Measured using the Self-Management Ability Scale-30 item questionnaire to assess ability and function. The SMAS consists of 30 items on four- and five-point Likert scales. Total score ranging from 0 to 100 with higher score indicating a higher function and ability, better outcome.
Time Frame: baseline; 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice
Number analyzed (Participants) | 80 | 91
score on a scale | 1.9 [-0.22 to 4.01] | 3.34 [1.72 to 4.97]

7. Secondary Outcome: Change in Daily Step Count
Description: Participants wore an Actigraph Activity Monitor for one week to measure daily steps.
Time Frame: baseline; 3 months
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice
Number analyzed (Participants) | 76 | 81
steps per day | 398.37 [-87.07 to 883.82] | 362.9 [-140.96 to 866.77]

8. Secondary Outcome: Change in Daily Total Physical Activity and Sedentary Time
Description: Participants wore an Actigraph Activity Monitor for one week to measure daily time spent doing sedentary (low energy expenditure) and non-sedentary (high energy expenditure) activities.
Time Frame: Baseline; 3 months
Population: For the interpretation of activity: a negative number in sedentary time and a positive number for overall physical activity are the goals (no defined minimal important difference)
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice
Number analyzed (Participants) | 76 | 81
minutes per day
  Average Daily Sedentary Time | 3.39 [-35.16 to 41.94] | -20.93 [-58.57 to 16.7]
  Average Daily Non-Sedentary Time | 1.14 [-28.39 to 30.66] | 9.34 [-16.82 to 35.51]

9. Secondary Outcome: Change in Duke-UNC Functional Social Support Questionnaire (FSSQ) Score
Description: The Duke-UNC Functional Social Support Questionnaire is an 8-item questionnaire that measures the amount of social support and availability of help from family and friends. The answers range from 1 "Much less than I would like" to 5 " As much as I would like". The scores from all 8 questions are summed (maximum 40) and then divided by 8 to get an average score. The higher the average score, the greater the perceived social support.
Time Frame: baseline; 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice
Number analyzed (Participants) | 95 | 102
score on a scale | -0.32 [-0.63 to 0] | -0.2 [-0.47 to 0.07]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 1 year.
Description: Adverse events were collected through follow up telephone calls with the subjects.
Arm/Group | Intervention- Home Pulmonary Rehabilitation | Control- Choice
All-Cause Mortality (participants affected / at risk) | 8/147 | 9/147
Serious Adverse Events (participants affected / at risk) | 2/147 | 1/147
Other Adverse Events (participants affected / at risk) | 0/147 | 1/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention- Home Pulmonary Rehabilitation (N=147) | Control- Choice (N=147)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Congestive Heart Failure Exacerbation (Cardiac disorders) | 1 | 0
Back Fractures (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention- Home Pulmonary Rehabilitation (N=147) | Control- Choice (N=147)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT04521608/Prot_SAP_000.pdf